CLINICAL TRIAL: NCT04670809
Title: A Randomized, Single Blind, Positive Parallel Controlled, Multicenter, Phase III Clinical Trial of Clevidipine Butyrate Injection in the Treatment of Hypertensive Emergencies
Brief Title: Safety and Efficacy Study of Clevidipine Butyrate Injection in Hypertensive Emergencies
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Yoko Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NJYK-LVDP-III
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hypertensive Emergency
MeSH Terms: conditions — Hypertensive Crisis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clevidipine Butyrate Injection (Experimental)
  Interventions: Drug: Clevidipine Butyrate Injection
- Ncardipine Hydrochloride Injection (Active Comparator)
  Interventions: Drug: Ncardipine Hydrochloride Injection

INTERVENTIONS:
Drug: Clevidipine Butyrate Injection — Initiate the intravenous infusion of Clevidipine Butyrate Injection at 2 mg/hour. The dose should be doubled every 3 minutes in the first 30 minutes if the desired blood pressure reduction (≥15% and ≤25%) is not achieved and the maximum dose is 32 mg/hour. The infusion duration should be at least 12 hours and less than 72 hours. Oral antihypertensive drugs should be given at about 2 hours before stopping infusion.
  Arms: Clevidipine Butyrate Injection
Drug: Ncardipine Hydrochloride Injection — Dilute the Ncardipine Hydrochloride Injection to 0.1mg/ml. Initiate the intravenous infusion at 0.5μg/(kg•min). A 0.5-1μg/(kg•min) dose should be added every 3 minutes in the first 30 minutes if the desired blood pressure reduction (≥15% and ≤25%) is not achieved and the maximum dose is 6μg/(kg•min). The infusion duration should be at least 12 hours and less than 72 hours. Oral antihypertensive drugs should be given at about 2 hours before stopping infusion.
  Arms: Ncardipine Hydrochloride Injection

SUMMARY:
The purpose of this study was to determine the efficacy and safety of clevidipine for treating Hypertensive emergencies（defined as systolic blood pressure >180 mmHg and/or diastolic blood pressure >120 mmHg, accompanied by acute organ damage）.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75, regardless of gender.
2. Blood pressure increased seriously in a short time, systolic blood pressure (SBP) > 180 mmHg and (or) diastolic blood pressure (DBP) > 120 mmHg (measured at an interval of 5 minutes, both blood pressure values should be > 180 / 120 mmHg), accompanied with progressive target organ damages as below or evidences of other target organ damage can be confirmed:

   * Hypertensive encephalopathy: headache, dizziness, irritability, nausea, vomiting, blurred vision and other symptoms;
   * Acute left heart failure: dyspnea, pulmonary rales, edema and other symptoms;
   * Unstable angina pectoris: ischemic chest pain with ST-T dynamic changes. Patients with SBP ≥ 220mmhg and / or DBP ≥ 140mmHg should be considered as hypertensive emergency;
3. The legal representative and / or patient agree to participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Patients with arterial dissection, acute hemorrhagic or ischemic stroke, and acute coronary syndrome in urgent need of surgical or emergency intervention;
2. Patients with severe aortic stenosis or severe mitral stenosis;
3. Patients with obstructive hypertrophic cardiomyopathy;
4. Patients who have used other intravenous antihypertensive drugs within 2 hours before entering this study;
5. Patients known to be intolerant or allergic to calcium channel blockers, or allergic to test drug ingredients, or allergic to soy / soy products or egg / egg products;
6. Patients with lipid metabolism defects, such as pathological hyperlipidemia, lipid nephropathy, or acute pancreatitis with hyperlipidemia;
7. Combined with other serious organ injury or serious complications which may affect the life of the subjects;
8. Patients with a history of mental illness;
9. Patients with known history of alcohol / drug abuse;
10. Those who have participated in other clinical trials and used test drugs 3 months before the trial;
11. Pregnant and lactating women;
12. Researchers do not consider it appropriate to participate in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Target reaching rate within 30 min | 30 min
  Proportion of subjects whose systolic blood pressure dropped to the target range (decrease ≥ 15% and ≤ 25% from baseline) in the first 30 minutes of administration.

SECONDARY OUTCOMES:
Mean time of target reaching | Procedure (whole infusion duration)
  Mean time for subjects to reach target systolic blood pressure.
Rate of successful conversion to oral antihypertensive drugs | 6 hours after intravenous administration
  Proportion of subjects who successfully converted to oral antihypertensive drugs within 6 hours after intravenous administration.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Anzhen Hospital，Capital Medical University, Beijing
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing

REFERENCES:
- [Derived] Lv Q, Chen C, Lin L, Zhao X, Chen J, Liang Z, Chai Y, Du B, Sun L, Chen X, Liu M, Zhang X, Cao Z, Zhang H, Chen D, Wang Z, Zhong Y, Zhu J, Gao F, Wang X, Zhang G, Li L, Ma J, Zhao M, Ouyang Y, Guo S, Wang H, Yang P, He R, Zhao Z, Sun L, Wu L, Wu Y, Liu X, Xu T, Li N, Zhu T, Ma C. Efficacy and safety of clevidipine emulsion injection compared with nicardipine in patients with hypertensive emergencies: a randomized, single-blind, positive-parallel-controlled, phase III clinical trial. J Hypertens. 2026 Jan 1;44(1):204-210. doi: 10.1097/HJH.0000000000004180. Epub 2025 Oct 23. PMID 41231022